CLINICAL TRIAL: NCT00271869
Title: Phase II Study for Treatment of Chronic Graft-Versus-Host Disease of the Liver or Lungs With Adjunct Extracorporeal Photoimmunotherapy
Brief Title: Treatment of Chronic GVHD of Liver or Lungs by ECP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK Nr. 368/2005
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2006-01-04 (Estimated); Status verified 2005-12

CONDITIONS: Chronic Graft-Versus Host Disease
Keywords: hematopoietic stem cell transplantation; graft-versus-host disease; treatment
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease

INTERVENTIONS:
Procedure: Extracorporeal photoimmunotherapy

SUMMARY:
Chronic graft-versus-host disease (GVHD) is a major complication of allogeneic hematopoietic stem cell transplantation and the leading cause of death more than 2 years after transplantation.During the past 30 years survival of patients with chronic GVHD has not improved and steroids remained the most often used therapy. Extracorporeal photoimmunotherapy (ECP)has shown to be efficacious in patients with GVHD. We propose a phase II study to evaluate the safety and efficacy of ECP as adjunct first-line therapy in patients with newly diagnosed chronic GVHD of liver or lungs and need for systemic immunosuppression defined according to the NIH consensus criteria.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one diagnostic clinical sign of chronic GVHD or an appropriate constellation of distinctive signs confirmed by biopsy or other relevant diagnostic tests
* Presence of liver or lung manifestations of chronic GVHD
* Indication for systemic immunosuppressive therapy defined according to NIH consensus
* No prior immunosuppressive therapy for chronic GVHD of the liver or lungs
* Adequate renal, hepatic, pulmonary and cardiac function
* Karnofsky performance score >- 50%
* Women of childbearing potential must agree to use a reliable method of birth control for the duration of the study
* Signed written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-12

PRIMARY OUTCOMES:
GVHD response of the liver or lungs

SECONDARY OUTCOMES:
transplant-related mortality
relapse-free survival
overall survival
time to complete resolution of chronic GVHD to first-line immunosuppressive therapy
time to discontinuation of immunosuppressive therapy
duration of response to first-line immunosuppressive therapy
percentage of patients in need of secondary treatment for chronic GVHD
incidence of bacterial, viral and fungal infections
side effects of ECP

CONTACTS AND LOCATIONS:
Overall Officials: Hildegard T Greinix, Professor of Medicine, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Medicine I, BMT, Vienna, Austria